CLINICAL TRIAL: NCT00287586
Title: Effects of Testosterone Replacement on Atherosclerosis Progression in Older Men With Low Testosterone Levels
Brief Title: Testosterone Replacement in Older Men and Atherosclerosis Progression
Acronym: TEAAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-24192
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Hypogonadism; Atherosclerosis
Keywords: Testosterone Replacement; Heart Disease; Vascular Disease; Risk Factors for Cardiovascular Disease; Cholesterol; Obesity; Blood pressure; Quality of Life
MeSH Terms: conditions — Hypogonadism; Atherosclerosis; Heart Diseases; Vascular Diseases; Obesity | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Testosterone (Active Comparator): Participants received 7.5 g of 1% testosterone gel to achieve a nominal delivery of 75 mg testosterone daily for 3 years. Dose adjustments were made by an unblinded observer. (Serum testosterone level measured on treatment day 15 was measured in a sample sent separately to the laboratory such that the results were reported directly to unblinded physician, who then communicated the decision about dose adjustment (or not) directly to the research pharmacist through e-mail.)
  Interventions: Drug: Testosterone Gel (Androgel)
- Placebo (Placebo Comparator): Participants received placebo-matching testosterone gel daily for 3 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Gel (Androgel) — 7.5 g of 1% testosterone gel to achieve a nominal delivery of 75 mg testosterone daily for 3 years
  Arms: Testosterone
Drug: Placebo — Placebo-matching testosterone gel daily for 3 years
  Arms: Placebo

SUMMARY:
As men grow older, their testosterone levels decrease with age. One-third of men, 70 years of age or older, have low testosterone levels. It is known that short-term testosterone replacement is safe, and can increase muscle strength and physical function, but the risks of long-term testosterone replacement in older men with low testosterone levels are incompletely understood.

Atherosclerosis is characterized by thickening of the artery walls, and the narrowing of the blood vessels as cholesterol is deposited in the lining of the arteries. It is the major cause of cardiovascular disease including ischemic heart disease (heart attacks) and stroke. Although, historically, there has been a widespread perception that higher levels of testosterone might increase the risk of atherosclerosis, the evidence from research does not support this. In observational studies, higher testosterone levels have been correlated with more favorable cardiovascular risk factors, and supplementation with testosterone to bring older men into the normal range for healthy younger men appears to improve several cardiovascular risk factors, and may slow the progression of atherosclerosis.

The primary purpose of this study is to look at the effects of testosterone replacement on the progression of atherosclerosis in older men. This study is also being done to find out whether replacement with testosterone in older men with low testosterone levels improves their health-related quality of life.

DETAILED DESCRIPTION:
Although short-term administration of testosterone in replacement doses is relatively safe, the risks of long-term testosterone administration in older men remain poorly understood. The two major areas of concern include the potential for increased risk of atherosclerotic heart disease and exacerbation of a pre-existing, subclinical prostate cancer. There is a widespread perception that testosterone supplementation adversely affects plasma lipoprotein profile and increases the risk of atherosclerotic heart disease; this premise is not supported by data. Thus, the long-term consequences of testosterone supplementation on the risk of atherosclerosis progression remain unknown. While supraphysiological doses of testosterone and non-aromatizable androgens frequently employed by body-builders undoubtedly decrease plasma high density lipoprotein (HDL)-cholesterol levels, physiologic testosterone replacement in older men has been associated with only a modest or no decrease in plasma HDL-cholesterol. Cross-sectional studies of middle-aged men find a direct, rather than an inverse, relationship between serum testosterone levels and plasma HDL-cholesterol concentrations as well as an inverse correlation between serum testosterone levels and visceral fat volume. Testosterone supplementation of middle-aged men with truncal obesity is associated with a reduction in visceral fat volume, serum glucose concentration, blood pressure, and an improvement in insulin sensitivity. All of these changes are associated with lower risk for atherosclerosis. These data suggest that serum testosterone levels in the range that is mid-normal for healthy young men are consistent with an optimal cardiovascular risk profile at any age, and that testosterone concentrations either above or below the physiologic male range may increase the risk of atherosclerotic heart disease. Studies in a low density lipoprotein (LDL)-receptor deficient mice provide compelling evidence that testosterone retards early atherogenesis, and that testosterone effects on atherogenesis are mediated through its conversion to estradiol by the action of aromatase enzyme that is expressed in the vessel wall. The effects of testosterone replacement on cardiovascular risk in humans have never been directly examined. Therefore, the primary objective of this study is to examine directly the effects of testosterone replacement on atherosclerosis progression in men by measuring common carotid artery intima-media thickness (CCA IMT) and coronary artery calcification (CAC) by multidetector computed tomography (MDCT), two independent measurements of generalized atherosclerosis.

The second objective of this study is to determine whether physiologic testosterone replacement of older men with low testosterone levels improves health-related quality of life. Aging-associated decline in physical, sexual, and cognitive functions contributes to diminished quality of life in older men. Although the pathophysiology of impairment in each of these subdomains of health-related quality of life is complex and multifactorial, one correctable cause of the diminished quality of life in older men is the decrease in serum testosterone concentrations. Total and free testosterone (T) levels decline with advancing age in normal men, with a significant number of men meeting usual criteria for hypogonadism by the sixth to seventh decades. Spontaneous and experimentally-induced androgen-deficiency in young men is associated with decreased muscle mass and strength and impaired sexual function. Because loss of muscle mass and function contributes to diminished health-related quality of life (HRQOL) in older men, anabolic therapies such as testosterone that increase muscle mass and strength, would be expected to improve physical function. In older men with low testosterone levels, testosterone might also improve sexual function and marital interaction. A growing body of literature suggests that testosterone impacts neuronal functioning and may affect cognitive performance. Because physical, sexual, and cognitive functions are important determinants of health-related quality of life, testosterone replacement of older men with low testosterone levels would be expected to improve general health perceptions.

The aging of humans is a recent evolutionary event. Of the thousand generations of men and women who have lived on this planet, only the humans of the last two generations could have hoped to live past the age of 50. The population is getting proportionally older. The number of people 85 years of age and older today is substantially greater than at the beginning of the 20th century. Advancing age is associated with decreased muscle mass and strength, and impairment of physical, sexual, and cognitive functions. Diminished muscle mass and strength increases the risk of falls, disability and poor quality of life. Age-related impairment of sexual and cognitive functions also contributes to overall reduction in quality of life. Testosterone replacement, by improving some aspects of physical, sexual and cognitive functions, would be expected to improve health-related quality of life.

Previous studies have established that testosterone replacement in older men with low testosterone levels increases muscle mass and strength. However, lack of information in two areas has prevented formulation of general recommendations about wider use of testosterone replacement in older men. First, the effectiveness of testosterone in improving physical function, quality of life, and other health-related outcomes has not been demonstrated. Second, while there is agreement that short-term administration of testosterone in replacement doses is safe, the long-term risks of testosterone supplementation in older men remain unknown. The areas of major concern are the risks of prostate cancer and heart disease. Because of the high prevalence, even small increases in the incidence rates of atherosclerotic heart disease associated with testosterone supplementation will have significant impact on overall morbidity and mortality, and health care costs. The study will evaluate one important aspect of the long-term safety of testosterone administration by directly examining its effects on the rate of progression of atherosclerosis. If the study demonstrates that testosterone retards atherosclerosis progression, then that would provide one additional reason for testosterone supplementation of older men with low testosterone levels. If the study demonstrates a neutral effect of testosterone on atherosclerosis progression, that information would also be reassuring and useful to regulatory agencies. This study will establish the efficacy of testosterone replacement in improving physical, sexual and cognitive functions that are major determinants of health-related quality of life in older men.

In spite of the paucity of efficacy and safety data, the sales of testosterone and other androgenic products have witnessed explosive growth because of increased media attention and public interest. During the summer of 2000, testosterone-related stories were on the cover of Time, Newsweek, New York Times, and Los Angeles Times. The prescription sales of testosterone that had been growing at 25-30% annual rate since 1993, almost doubled in the year 2000, and have cumulatively increased 500% since 1993 (Source: IMS Sales Data, provided by Reed Selby, Marketing Director for ALZA Corporation). The growing testosterone use in older men, without a clear understanding of its benefits or long-term risks, has raised concern among regulatory agencies. The proposed study by providing definitive information on the effects of testosterone replacement on several measures of efficacy and safety in older men would facilitate an analysis of its risk:benefit ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or greater
* Hypogonadism, Testosterone 100-400 ng/dl or Free Testosterone < 50 pg/ml
* Generally good health
* At least 8 years of primary school education
* Able to pass screening test for dementia
* Able to give informed consent

Exclusion Criteria:

* Testosterone level < 100 ng/dl (these individuals will be referred for evaluation of severe hypogonadism)
* Use of testosterone or other androgens [dehydroepiandrosterone (DHEA), Androstenedione] in last year
* Use of growth hormone in the last year
* Current alcohol of drug dependence [Alcohol Use Disorders Identification Test (AUDIT) Score > 8]
* Diseases known to affect gonadal function
* Medications known to affect gonadal function eg. anticonvulsants, glucocorticoids such as prednisone
* Prostate cancer, breast cancer
* Any cancer that may limit life expectancy to less than 5 years
* Limiting neuromuscular, joint or bone disease
* History of stroke with residual neurologic deficit
* Neurologic condition that would impair cognitive function including:

epilepsy, multiple sclerosis, human immunodeficiency virus (HIV), Parkinson's disease, stroke

* Psychiatric disorder in the last year meeting Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSMIV) Axis 1 criteria
* Use of psychotropic medicine for at least 6 months
* Dementia as assessed by (Telephone Interview for Cognitive Status modified score less than 31)
* Severe symptoms of benign prostatic hyperplasia (BPH) (American Urological Association symptom index score greater than 21)
* Prostate nodule or induration of digital rectal exam (DRE)
* Prostate specific antigen (PSA) greater than 4 unless participant has had a negative transrectal biopsy within last 3 months
* Limiting heart disease in including New York (NY) Class III or IV - congestive heart failure, unstable angina, or myocardial infarction (MI) in last 3 months
* Liver function tests [aspartate aminotransferase (AST) and alanine aminotransferase(ALT)] greater than 3 times the upper limit of the reference range
* Serum creatinine (Cr) greater than 2.5 mg/dl
* Hematocrit greater than 48%
* Hemoglobin (Hb)A1c greater than 9.0%
* Untreated thyroid disease
* Uncontrolled hypertension (systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg)
* Body mass index (BMI greater than 35 kg/m2)
* Untreated severe obstructive sleep apnea
* Development of electrocardiogram (EKG) changes consistent with myocardial ischemia or changes in blood pressure during cardiopulmonary exercise testing will be excluded from testing of muscle strength and physical function.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2012-02-07 (Actual); Study Completion 2012-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Boston University / Boston Medical Center, Boston, MA
Locations (3):
- United States (3):
  - Kronos Longevity Research Institute, Phoenix, Arizona
  - Charles R. Drew University of Medicine and Science, Los Angeles, California
  - Boston University / Boston Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Huang G, Pencina KM, Li Z, Basaria S, Bhasin S, Travison TG, Storer TW, Harman SM, Tsitouras P. Long-Term Testosterone Administration on Insulin Sensitivity in Older Men With Low or Low-Normal Testosterone Levels. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1678-1685. doi: 10.1210/jc.2017-02545. PMID 29373734
- [Derived] Bhasin S, Travison TG, O'Brien L, MacKrell J, Krishnan V, Ouyang H, Pencina K, Basaria S. Contributors to the substantial variation in on-treatment testosterone levels in men receiving transdermal testosterone gels in randomized trials. Andrology. 2018 Jan;6(1):151-157. doi: 10.1111/andr.12428. Epub 2017 Oct 5. PMID 28981994
- [Derived] Gagliano-Juca T, Icli TB, Pencina KM, Li Z, Tapper J, Huang G, Travison TG, Tsitouras P, Harman SM, Storer TW, Bhasin S, Basaria S. Effects of Testosterone Replacement on Electrocardiographic Parameters in Men: Findings From Two Randomized Trials. J Clin Endocrinol Metab. 2017 May 1;102(5):1478-1485. doi: 10.1210/jc.2016-3669. PMID 27992261
- [Derived] Storer TW, Basaria S, Traustadottir T, Harman SM, Pencina K, Li Z, Travison TG, Miciek R, Tsitouras P, Hally K, Huang G, Bhasin S. Effects of Testosterone Supplementation for 3 Years on Muscle Performance and Physical Function in Older Men. J Clin Endocrinol Metab. 2017 Feb 1;102(2):583-593. doi: 10.1210/jc.2016-2771. PMID 27754805
- [Derived] Huang G, Wharton W, Bhasin S, Harman SM, Pencina KM, Tsitouras P, Li Z, Hally KA, Asthana S, Storer TW, Basaria S. Effects of long-term testosterone administration on cognition in older men with low or low-to-normal testosterone concentrations: a prespecified secondary analysis of data from the randomised, double-blind, placebo-controlled TEAAM trial. Lancet Diabetes Endocrinol. 2016 Aug;4(8):657-665. doi: 10.1016/S2213-8587(16)30102-4. Epub 2016 Jul 1. PMID 27377542
- [Derived] Basaria S, Harman SM, Travison TG, Hodis H, Tsitouras P, Budoff M, Pencina KM, Vita J, Dzekov C, Mazer NA, Coviello AD, Knapp PE, Hally K, Pinjic E, Yan M, Storer TW, Bhasin S. Effects of Testosterone Administration for 3 Years on Subclinical Atherosclerosis Progression in Older Men With Low or Low-Normal Testosterone Levels: A Randomized Clinical Trial. JAMA. 2015 Aug 11;314(6):570-81. doi: 10.1001/jama.2015.8881. PMID 26262795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 156 | 152
Intent-to-treat: Received Study Drug | 155 | 151
Completed | 111 | 100
Not Completed | 45 | 52
Not completed — Withdrew Consent | 19 | 30
Not completed — Lost to Follow-up | 5 | 4
Not completed — Death | 2 | 3
Not completed — Elevated Hematocrit | 3 | 0
Not completed — Rash | 3 | 0
Not completed — Elevated Prostate Specific Antigen | 2 | 0
Not completed — Stroke | 2 | 0
Not completed — Myocardial Infarction | 1 | 0
Not completed — Lower Urinary Tract Symptoms | 1 | 0
Not completed — Cognitive Impairment | 1 | 0
Not completed — Pancreatic Cancer | 1 | 3
Not completed — Sleep Apnea | 1 | 0
Not completed — Shoulder Pain | 1 | 0
Not completed — Inappropriate Behaviour with Staff | 1 | 0
Not completed — Nonadherence | 1 | 1
Not completed — Enrolled in Another Study | 1 | 0
Not completed — Major Depression | 0 | 2
Not completed — Lung Cancer | 0 | 2
Not completed — Elevated IPSS Score | 0 | 1
Not completed — Retroperitoneal Cancer | 0 | 1
Not completed — Mastodynia and Gynecomastia | 0 | 1
Not completed — Mood Swings and Irritability | 0 | 1
Not completed — Bradycardia | 0 | 1
Not completed — Itchy Swollen Eyes | 0 | 1
Not completed — Recurrent Melanoma | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 155 | 151 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (5.0) | 68.3 (5.3) | 67.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 155 | 151 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Common Carotid Artery Intima-Media Thickness (IMT)
Description: B-mode carotid artery images for IMT were acquired from the far wall of the distal centimeter of the right carotid artery with high-resolution ultrasound equipment. IMT is used as a predictor of the incidence of cardiovascular events. An increase in the IMT thickness is associated with a higher incidence of cardiovascular events. Less thickening is best. Change is expressed in millimeters (mm).
Time Frame: Baseline and Month 36
Population: All participants from the Intent-to-treat population, all randomized and treated participants, with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 155 | 151
mm
  Baseline | 0.877 (0.210) | 0.879 (0.199)
  Change at Month 36: number analyzed (Participants) | 101 | 92
  Change at Month 36 | 0.036 (0.059) | 0.033 (0.077)

2. Primary Outcome: Change From Baseline in Coronary Artery Calcium Score
Description: A multiple detector computed tomography (MDCT) scan was performed. Proximal coronary arteries were visualized, and at least 30 consecutive images were obtained at 3-mm intervals. Coronary calcium was defined as a plaque of at least 3 contiguous pixels (area, 1.02 mm^2) with a density of more than 130 Hounsfield units.The lesion score was calculated by multiplying lesion area by a density factor derived from Hounsfield units. The Agatston method was used to determine the total calcium score by summing the lesion scores from the left main, left anterior descending, circumflex, and right coronary arteries. The Agatston score is the measure of calcification in arteries expressed on continuous scale with "0" value (better) indicating no calcification and score above 400 (worse) indicating high calcification. There is no upper limit for this measure. A positive change from baseline indicates a worsening.
Time Frame: Baseline and Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 155 | 151
score on a scale
  Baseline: number analyzed (Participants) | 140 | 132
  Baseline | 451.78 (715.41) | 508.31 (694.87)
  Change at Month 36: number analyzed (Participants) | 92 | 92
  Change at Month 36 | 103.61 (289.45) | 124.54 (208.42)

3. Secondary Outcome: Change From Baseline in Lipid Profiles
Description: Laboratory tests included in the lipid profile were Total Cholesterol, High Density Lipoprotein-Cholesterol (HDL-C), Low Density Lipoprotein-Cholesterol (LDL-C) and Triglycerides.Lower values for Total Cholesterol, LDL-C are better and a negative change from Baseline indicates improvement. Higher values for HDL-C are better and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 155 | 151
mg/dL
  Total Cholesterol, Baseline: number analyzed (Participants) | 153 | 147
  Total Cholesterol, Baseline | 187.15 (42.09) | 183.44 (36.68)
  Total Cholesterol, Change at Month 36: number analyzed (Participants) | 101 | 96
  Total Cholesterol, Change at Month 36 | -14.88 (35.92) | -12.56 (33.90)
  HDL-C, Baseline: number analyzed (Participants) | 152 | 146
  HDL-C, Baseline | 47.11 (11.97) | 48.71 (14.21)
  HDL-C, Change at Month 36: number analyzed (Participants) | 100 | 95
  HDL-C, Change at Month 36 | 0.18 (9.69) | 2.00 (11.08)
  LDL-C, Baseline: number analyzed (Participants) | 151 | 146
  LDL-C, Baseline | 115.64 (35.18) | 109.66 (31.86)
  LDL-C, Change at Month 36: number analyzed (Participants) | 99 | 95
  LDL-C, Change at Month 36 | -11.24 (26.80) | -13.92 (30.80)
  Triglycerides, Baseline: number analyzed (Participants) | 154 | 146
  Triglycerides, Baseline | 142.695 (87.93) | 138.95 (76.37)
  Triglycerides, Change at Month 36: number analyzed (Participants) | 101 | 95
  Triglycerides, Change at Month 36 | -19.41 (73.69) | -12.62 (84.62)

4. Secondary Outcome: Changes in Biomarkers of Inflammation
Time Frame: Three years
Population: No analysis was performed. No funds were left to cover the costs of the assays for inflammation biomarkers.
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Blood Pressure
Time Frame: Three years
Population: No analysis was performed. Although blood pressure measurements were standardized within a trial site, there is a possibility that measurement techniques might have varied across the three trial sites over the trial's long duration. For this reason we decided not to include blood pressure data in the results.
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Complex Figure (Immediate) and Complex Figure (Delayed)
Description: Cognitive Function was assessed by Complex Figure (Immediate) and (Delayed). The Complex Figure Test consists of three tasks: copy, immediate recall, and delayed recall. Participants were presented with a complex design and then asked to draw the same figure. Subsequently, they were instructed to draw what they remembered immediately, and after a 30 minute delay. Scoring was based on the number of correct items for a total possible score of 0 (worst) to 36 (Best). A positive change from Baseline indicates improvement. A negative change from Baseline indicates a worsening.
Time Frame: Baseline and Month 36
Population: All participants from the Intent-to-treat population, all randomized and treated participants, with cognitive baseline data and data available at the given time-point.
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
correct items
  Complex Figure:Immediate, Baseline: number analyzed (Participants) | 124 | 124
  Complex Figure:Immediate, Baseline | 20.95 (6.50) | 20.31 (6.20)
  Complex Figure:Immediate, Change at Month 36: number analyzed (Participants) | 84 | 79
  Complex Figure:Immediate, Change at Month 36 | -1.25 (4.90) | -0.24 (6.11)
  Complex Figure:Delayed, Baseline: number analyzed (Participants) | 121 | 124
  Complex Figure:Delayed, Baseline | 20.28 (6.08) | 19.75 (6.11)
  Complex Figure:Delayed, Change at Month 36: number analyzed (Participants) | 82 | 77
  Complex Figure:Delayed, Change at Month 36 | -0.49 (5.20) | -0.24 (5.74)

7. Secondary Outcome: Change From Baseline in Paragraph Recall Test (Delayed)
Description: Cognitive Function was assessed by the Paragraph Recall Test (Delayed). In the Paragraph Recall Test, participants were read two short paragraphs and asked to recall them immediately and after a 30 minute delay, using the exact words that were read aloud. Scoring was based on the number of items correctly recalled. More items correctly recalled is best and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
correct items
  Paragraph: Delayed, Baseline: number analyzed (Participants) | 139 | 139
  Paragraph: Delayed, Baseline | 13.69 (6.37) | 13.57 (6.12)
  Paragraph:Delayed, Change at Month 36: number analyzed (Participants) | 92 | 88
  Paragraph:Delayed, Change at Month 36 | 2.15 (6.05) | 1.72 (4.82)

8. Secondary Outcome: Change From Baseline in the Buschke Selective Reminding Test (Delayed)
Description: Cognitive function was assessed by the Buschke Selective Reminding Test. In the Buschke Selective Reminding Test, participants were read 12 words and asked to recall as many words as possible. Subsequent trials included only those words that were not recalled in the preceding trial. Individuals were also asked to recall the list 30 minutes later. To assess phonemic and category fluency, participants were asked to name as many items from a given category as possible in 1 minute. Higher number of correct items is best and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
correct items
  Buschke Total Correct Delayed, Baseline: number analyzed (Participants) | 138 | 137
  Buschke Total Correct Delayed, Baseline | 8.00 (2.80) | 7.76 (2.69)
  Buschke Total Correct Delayed, Change at Month 36: number analyzed (Participants) | 96 | 92
  Buschke Total Correct Delayed, Change at Month 36 | 0.47 (2.46) | 0.85 (2.21)

9. Secondary Outcome: Change From Baseline in the Verbal Fluency Test
Description: Cognitive function was assessed by the Verbal Fluency Test. Participants were asked to name as many letters from a given category as possible in 1 minute. Higher number of letters is best and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
letters
  Baseline: number analyzed (Participants) | 137 | 139
  Baseline | 26.96 (10.25) | 27.02 (8.97)
  Change at Month 36: number analyzed (Participants) | 96 | 93
  Change at Month 36 | 2.86 (8.84) | 1.77 (7.35)

10. Secondary Outcome: Change From Baseline in the Category Fluency Test
Description: Cognitive function was assessed by the Category Fluency Test. Participants were asked to name as many items from a given category as possible. Higher number of items named is best and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: items
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
items
  Category Fluency, Baseline: number analyzed (Participants) | 135 | 138
  Category Fluency, Baseline | 18.07 (5.61) | 18.01 (5.62)
  Category Fluency, Change at Month 36: number analyzed (Participants) | 95 | 93
  Category Fluency, Change at Month 36 | 2.25 (6.81) | 0.37 (6.77)

11. Secondary Outcome: Change From Baseline in the Stroop Interference Test
Description: Cognitive function was assessed by the Stroop Interference Test. In the Stroop Interference Test, participants were presented with a word list of colors printed in ink of a color different from how the printed word read. Participants were instructed to read aloud the color of the ink in which a word was printed, while not verbalizing the word itself. The time in seconds that the items were correctly identified was recorded. Less time is better and a negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
seconds
  Stroop Interference, Baseline: number analyzed (Participants) | 137 | 140
  Stroop Interference, Baseline | 55.64 (15.60) | 56.84 (15.85)
  Stroop Interference, Change at Month 36: number analyzed (Participants) | 95 | 93
  Stroop Interference, Change at Month 36 | -1.07 (14.48) | 0.99 (16.10)

12. Secondary Outcome: Change From Baseline in the Trail Making Test B
Description: Cognitive function was assessed by the Trail Making Test B. Trail Making Test B involved participants connecting numbers (1-13) and letters (A-L) alternately (1-A, 2-B, etc) on a piece of paper as quickly as possible. Scores represent the time it takes the participant to complete the test. Less time is best and a negative change from Baseline indicates improvement. A positive change from Baseline indicates a worsening.
Time Frame: Baseline and Month 36
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 140 | 140
seconds
  Trails B, Baseline: number analyzed (Participants) | 135 | 131
  Trails B, Baseline | 98.52 (42.40) | 97.57 (31.82)
  Trails B, Change at Month 36: number analyzed (Participants) | 82 | 81
  Trails B, Change at Month 36 | 3.88 (34.15) | 11.26 (40.61)

13. Secondary Outcome: Change From Baseline in Chest Press Strength and Leg Press Strength
Description: Maximal voluntary strength of the lower and upper extremities was assessed using the one repetition maximum (1-RM) method for the seated leg press and chest press exercises. Participants were positioned with standardized seat position and foot placement that allowed 90° of knee flexion for the leg press exercise. Seat height and handle position was standardized for the chest press. Participants were familiarized with the exercises, practiced the technique and completed a 5-minute warm-up. The 1-RM procedure consisted of a warm up set with 5 to 8 repetitions at a resistance set to about 50% of the participant's estimated 1-RM and progressed with increasing loads interspersed with standardized rest periods until the participant was able to perform only one full-range-of-motion repetition.
Time Frame: Baseline and Month 36
Population: All participants from the Intent-to-treat population, all randomized and treated participants, with baseline physical function data and data available at the given time-point.
Measure: Mean (Standard Deviation); unit: newton
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 135 | 121
newton
  Chest Press Strength, Baseline: number analyzed (Participants) | 125 | 110
  Chest Press Strength, Baseline | 516.99 (133.37) | 513.83 (104.92)
  Chest Press Strength, Change at Month 36: number analyzed (Participants) | 82 | 67
  Chest Press Strength, Change at Month 36 | -12.73 (54.20) | -26.20 (40.88)
  Leg Press Strength, Baseline: number analyzed (Participants) | 128 | 109
  Leg Press Strength, Baseline | 2270.37 (424.81) | 2233.74 (416.06)
  Leg Press Strength, Change at Month 36: number analyzed (Participants) | 84 | 68
  Leg Press Strength, Change at Month 36 | -37.26 (230.42) | -65.33 (251.94)

14. Secondary Outcome: Change From Baseline in Unloaded Stair Climb Power and Loaded Stair Climb Power
Description: Physical Function was evaluated using two tests of stair climb power using an indoor 12-step staircase. One test consisted of ascending the 12-steps as rapidly as possible without running (unloaded stair climb) while the second test required participants to carry a load equivalent to 20% of their baseline body weight evenly distributed in two canvas tote bags (loaded stair climb). Time to ascend the stairs was measured electronically with a digital clock and switch mats placed at the base of the steps and on the 12th step. Power in watts is calculated by the following: [body weight (kilograms) * distance (meters)/ (time/60)] /6.12. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 135 | 121
watts
  Unloaded Stair Climb Power, Baseline: number analyzed (Participants) | 116 | 98
  Unloaded Stair Climb Power, Baseline | 536.33 (134.40) | 535.78 (125.70)
  Unloaded Stair Climb Power, Change at Month 36: number analyzed (Participants) | 77 | 61
  Unloaded Stair Climb Power, Change at Month 36 | -8.17 (71.60) | -12.89 (64.28)
  Loaded Stair Climb Power, Baseline: number analyzed (Participants) | 106 | 89
  Loaded Stair Climb Power, Baseline | 581.24 (148.73) | 594.84 (150.28)
  Loaded Stair Climb Power, Change at Month 36: number analyzed (Participants) | 67 | 54
  Loaded Stair Climb Power, Change at Month 36 | -8.44 (70.56) | -12.76 (63.13)

15. Secondary Outcome: Change in Sexual Function as Assessed by the International Index of Erectile Function (IIEF)
Description: IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (6 questions), orgasmic function (2 questions), sexual desire (2 questions), intercourse satisfaction (3 questions), and overall sexual satisfaction (2 questions). Each question was answered on a 5-point scale from 1 to 5 (best) with a total possible score range of 0 to 75 with higher scores representing better function. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 155 | 151
score on a scale
  Erectile Function, Baseline: number analyzed (Participants) | 129 | 125
  Erectile Function, Baseline | 18.33 (10.11) | 18.67 (10.64)
  Erectile Function, Change at Month 36: number analyzed (Participants) | 104 | 94
  Erectile Function, Change at Month 36 | -0.15 (7.40) | -0.80 (7.55)
  Orgasmic Function, Baseline: number analyzed (Participants) | 134 | 126
  Orgasmic Function, Baseline | 7.37 (3.61) | 6.38 (3.86)
  Orgasmic Function, Change at Month 36: number analyzed (Participants) | 108 | 97
  Orgasmic Function, Change at Month 36 | -0.65 (3.35) | 0.24 (3.44)
  Sexual Desire, Baseline: number analyzed (Participants) | 133 | 125
  Sexual Desire, Baseline | 6.89 (2.04) | 6.58 (2.19)
  Sexual Desire, Change at Month 36: number analyzed (Participants) | 108 | 96
  Sexual Desire, Change at Month 36 | 0.18 (1.94) | 0.07 (1.87)
  Intercourse Satisfaction, Baseline: number analyzed (Participants) | 131 | 127
  Intercourse Satisfaction, Baseline | 8.32 (5.92) | 8.14 (5.94)
  Intercourse Satisfaction, Change at Month 36: number analyzed (Participants) | 105 | 97
  Intercourse Satisfaction, Change at Month 36 | 0.05 (4.56) | -0.71 (4.11)
  Overall Satisfaction, Baseline: number analyzed (Participants) | 123 | 116
  Overall Satisfaction, Baseline | 6.24 (2.84) | 6.12 (2.64)
  Overall Satisfaction, Change at Month 36: number analyzed (Participants) | 99 | 87
  Overall Satisfaction, Change at Month 36 | 0.40 (2.77) | 0.81 (2.54)
  Total Score, Baseline: number analyzed (Participants) | 117 | 110
  Total Score, Baseline | 48.48 (21.09) | 49.67 (23.25)
  Total Score, Change at Month 36: number analyzed (Participants) | 97 | 85
  Total Score, Change at Month 36 | 0.22 (15.54) | -0.39 (15.32)

16. Secondary Outcome: Change in Health Quality of Life (QoL) as Assessed by Short Form 36 (SF-36)
Description: The SF-36 measures 8 domains of the QoL: physical function, bodily pain, vitality, role limitations due to physical problems, general health perceptions, emotional well-being, social function, and role limitations due to emotional problems. Each domain is scored separately from 0 to 100 with higher scores representing better health-related QoL. The Overall Score is the average of the individual domain scores. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 155 | 151
score on a scale
  Energy/Fatigue, Baseline: number analyzed (Participants) | 60 | 58
  Energy/Fatigue, Baseline | 69.92 (18.47) | 71.21 (14.67)
  Energy/Fatigue, Change at Month 36: number analyzed (Participants) | 39 | 44
  Energy/Fatigue, Change at Month 36 | -1.45 (13.40) | -0.46 (12.57)
  Emotional Well-Being, Baseline: number analyzed (Participants) | 60 | 58
  Emotional Well-Being, Baseline | 82.67 (12.64) | 83.17 (11.38)
  Emotional Well-Being, Change at Month 36: number analyzed (Participants) | 39 | 44
  Emotional Well-Being, Change at Month 36 | -1.16 (14.76) | 0.91 (11.60)
  Role Limitations/Emotional Problems, Baseline: number analyzed (Participants) | 60 | 58
  Role Limitations/Emotional Problems, Baseline | 90.00 (23.21) | 89.08 (26.04)
  Role Limitations/Emotional Problems,Change: number analyzed (Participants) | 39 | 44
  Role Limitations/Emotional Problems,Change | 3.51 (32.69) | -9.09 (34.00)
  Social Functioning, Baseline: number analyzed (Participants) | 60 | 58
  Social Functioning, Baseline | 90.42 (16.17) | 92.89 (13.06)
  Social Functioning, Change at Month 36: number analyzed (Participants) | 39 | 44
  Social Functioning, Change at Month 36 | -3.29 (22.64) | -4.83 (14.06)
  Physical Functioning, Baseline: number analyzed (Participants) | 60 | 58
  Physical Functioning, Baseline | 82.00 (20.15) | 83.28 (18.79)
  Physical Functioning, Change at Month 36: number analyzed (Participants) | 39 | 44
  Physical Functioning, Change at Month 36 | -3.82 (21.20) | -2.39 (21.09)
  Role Limitations/Physical Health, Baseline: number analyzed (Participants) | 60 | 58
  Role Limitations/Physical Health, Baseline | 80.00 (30.81) | 88.79 (21.55)
  Role Limitations,/Physical Health, Change: number analyzed (Participants) | 39 | 44
  Role Limitations,/Physical Health, Change | -1.97 (24.23) | -9.66 (34.61)
  Pain, Baseline: number analyzed (Participants) | 60 | 58
  Pain, Baseline | 82.83 (17.29) | 82.24 (15.84)
  Pain, Change at Month 36: number analyzed (Participants) | 39 | 44
  Pain, Change at Month 36 | -7.96 (14.81) | -5.97 (17.90)
  General Health, Baseline: number analyzed (Participants) | 60 | 58
  General Health, Baseline | 74.17 (19.51) | 76.72 (15.18)
  General Health, Change at Month 36: number analyzed (Participants) | 39 | 44
  General Health, Change at Month 36 | -0.53 (11.90) | -3.75 (14.59)
  Overall Score, Baseline: number analyzed (Participants) | 60 | 58
  Overall Score, Baseline | 81.50 (14.12) | 83.42 (12.45)
  Overall Score, Change at Month 36: number analyzed (Participants) | 39 | 44
  Overall Score, Change at Month 36 | -2.08 (11.88) | -4.40 (12.24)

ADVERSE EVENTS:
Arm/Group | Testosterone | Placebo
Serious Adverse Events (participants affected / at risk) | 24/155 | 25/151
Other Adverse Events (participants affected / at risk) | 33/155 | 20/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=155) | Placebo (N=151)
Death (General disorders) | 1 | 6
Pulmonary carcinoma complications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Resulting in death
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Resulting in death
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Resulting in death
Angina pectoris (Cardiac disorders) | 1 | 3
Appendicitis (Infections and infestations) | 0 | 1
Appendectomy (Surgical and medical procedures) | 0 | 1
Bacterial septicemia (Infections and infestations) | 0 | 1
Triple by-pass surgery (Surgical and medical procedures) | 0 | 1
Coronary artery bypass graft (Surgical and medical procedures) | 0 | 1
Chest pain (General disorders) | 1 | 1
Colitis with abscess and fistula (Infections and infestations) | 0 | 1
Colonic diverticulitis (Gastrointestinal disorders) | 0 | 1
Complete ankle replacement surgery (Surgical and medical procedures) | 0 | 1
Congestive heart failure (Cardiac disorders) | 0 | 1
Congestive heart failure exacerbation (Cardiac disorders) | 0 | 1
Lung mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
E.coli infection (Infections and infestations) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningitis not otherwise specified (NOS) (Infections and infestations) | 0 | 1
Bacteriemia (Infections and infestations) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mugged (Injury, poisoning and procedural complications) | 0 | 1 — Resulted in death
Pulseless electrical activity (PEA) cardiac arrest (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Lung cancer reaccurence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung pulmonary nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Slient myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coronary angiogram resulted in 2 occluded vessels (Injury, poisoning and procedural complications) | 0 | 1
Coronary stent procedure (Surgical and medical procedures) | 1 | 1
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute posterior myocardial infarction (Cardiac disorders) | 1 | 0
Angioplasty (Surgical and medical procedures) | 2 | 0
Aspiration pneumonia (Infections and infestations) | 1 | 0
Bilateral toe gangrene (Infections and infestations) | 1 | 0
Cellulites on right foot and calf (Infections and infestations) | 1 | 0
Cerebellar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Elevated blood pressure (Investigations) | 1 | 0
Complete left knee replacement surgery (Surgical and medical procedures) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary heart disease (Cardiac disorders) | 1 | 0
Cerebrovascular accident (CVA) (Nervous system disorders) | 3 | 0
Exertional chest pains (General disorders) | 1 | 0
Herniated free fragment with right lumbar radiculopathy (Nervous system disorders) | 1 | 0
Leg pain (General disorders) | 1 | 0
Localized prostate adeno-carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Neoplasm left kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Saphenous vein graft occlusion (Vascular disorders) | 1 | 0
Pancreatic tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Quadruple by-pass surgery (Surgical and medical procedures) | 1 | 0
Right hemispheric subacute stroke (Nervous system disorders) | 1 | 0
Right knee re-placement surgery (Surgical and medical procedures) | 1 | 0
Second-degree atrioventricular heart block (Cardiac disorders) | 1 | 0
Dual chamber pace maker placement (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=155) | Placebo (N=151)
Elevated Prostate-Specific Antigen (PSA) (Investigations) | 16 | 9
Upper respiratory infection (Infections and infestations) | 12 | 12
Elevated hematocrit (HCT) (Investigations) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes